CLINICAL TRIAL: NCT00257491
Title: An Open-label Study to Evaluate the Trough and Peak Effect of Once Daily Micardis Plus (Telmisartan 80mg / Hydrochlorothiazide 12.5 mg) by 24 ABPM in Patients With Mild to Moderate Essential Hypertension
Brief Title: Study to Evaluate the Trough and Peak Effect of Once Daily Telmisartan 80 mg/Hydrochlorothiazide 12.5 mg (Micardis Plus) by Ambulatory Blood Pressure Monitoring (ABPM) in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 502.488
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

INTERVENTIONS:
Drug: Telmisartan
Drug: Telmisartan/HCTZ

SUMMARY:
To evaluate the trough and peak effect of once daily MICARDIS PLUS (Telmisartan 80 mg/hydrochlorothiazide 12.5 mg) by 24 ABPM in patients with mild to moderate essential hypertension.

DETAILED DESCRIPTION:
This study is designed as an open label study. After a 2-week placebo run-in phase, qualified patients will be administered with telmisartan 80mg for 2 weeks, then forcefully titrated to telmisartan 80 mg and hydrochlorothiazide 12.5 mg fixed dose combination for 6 weeks. 24 hour ABPM will be performed at the end of placebo run-in period (baseline) and after 8 weeks of active treatment.

Study Hypothesis:

The primary analyses will be the calculation of trough to peak ratios (T/P ratios) for DBP and SBP. The T/P ratio will be calculated on the basis of changes in hourly means (related to dosing time) from baseline (DeltaHM). Trough is defined as the mean of the last three hours of the 24-hour dosing interval. Peak is the greatest reduction in hourly means in hours 2 to 8 after dosing. Thus, T/P is calculated as T/P = mean(DeltaHM22 - DeltaHM24)/min (DeltaHM2 - DeltaHM8).

Comparison(s):

To assess trough/peak ratio of once daily Micardis plus by 24 ABPM in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. History of mild-to-moderate essential hypertension defined by a mean seated DBP >= 95 and <= 109 mmHg, and SBP < 180mmHg measured by manual cuff sphygmomanometer at visit 2.

   Note: The manual cuff value is calculated as the mean of three seated measurements collected 2 minutes apart, after the patient has been seated quietly for 5 minutes. For calculation of mean values by the investigator, decimal places should be rounded to integers as usual (e.g., a DBP of 94.7 would be rounded to 95 mmHg and a DBP of 109.3 would be rounded to 109 mmHg).
2. Participants between 18 and 80 years of age.
3. Ability to provide written informed consent. 4.24 hour mean DBP >= 85 mmHg at visit 3.

5.Ability to stop any current antihypertensive therapy without risk to the patient (investigators discretion).

Exclusion Criteria:

1. Patients taking more than three anti-hypertensive medications at the screening visit.
2. Pre-menopausal women (last menstruation <= 1 year prior to start of screening):

   * Who are not surgically sterile (hysterectomy, tubal ligation).
   * Who are NOT practicing acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the study. Acceptable methods of birth control include IUD, oral, implantable or injectable contraceptives.
3. Any woman:

   * Who has a positive urine pregnancy test at screening (Visit 1).
   * Who is nursing.
4. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   * SGPT(ALT) or SGOT(AST) greater than two times the upper limit of normal.
   * Serum creatinine > 3.0 mg/dL (or 265 mmol/L) or creatinine clearance < 0.6 ml/sec.
5. Clinically relevant hypokalaemia or hyperkalaemia.
6. Uncorrected volume depletion.
7. Uncorrected sodium depletion.
8. Hereditary fructose intolerance.
9. Biliary obstructive disorders, cholestasis or moderate to severe hepatic insufficiency.
10. Known or suspected secondary hypertension.
11. Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney.
12. Congestive heart failure (NYHA functional class CHF III-IV refer to Appendix 11. 1).
13. Unstable angina within the past three months.
14. Stroke within the past six months.
15. Myocardial infarction or cardiac surgery within the past three months.
16. PTCA within the past three months.
17. Patients who have previously experienced symptoms characteristic of angiodema during treatment with ACE inhibitor or angiotensin II receptor antagonists.
18. Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator.
19. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08

PRIMARY OUTCOMES:
To assess trough/peak ratio of once daily Micardis plus by 24 ABPM in patients with mild to moderate essential hypertension.

SECONDARY OUTCOMES:
Smooth Index for DBP and SBP Change from the baseline in the ABPM endpoint: 24 hour mean, daytime mean , nighttime mean, morning mean, last 6-hours of the dosing interval mean SBP, DBP,MAP and HR.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China